CLINICAL TRIAL: NCT00630617
Title: Project FAMILIA Giya Marianas: Childhood Obesity Prevention Program
Brief Title: Childhood Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Michigan University (Other)
Collaborators: Hillblom Foundation (Unknown); Commonwealth of the Northern Marianna Islands Public School System (Unknown)
Responsible Party: Mozhdeh B. Bruss, PhD, MPH, RD/Associate Professor, Western Michigan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-06-14
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Childhood Obesity; Diabetes
Keywords: Obesity; Prevention; Childhood; Children; Primary care-giver
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus; Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Diet, Physical activity, Physical inactivity — Community based participatory research design

SUMMARY:
To develop and evaluate a culturally appropriate childhood obesity prevention program targeting primary care-givers of third grade students. The cognitive-behavioral lifestyle intervention consisted of eight, 90-minute sessions at the elementary schools.

Primary outcome: body mass index of third graders and their primary care-givers Primary objective: To engage primary care-givers of third grand children in identifying and creating health promoting culturally appropriate environments for young children.

DETAILED DESCRIPTION:
The sessions include information about energy balance, portion control, appropriate amounts and types of physical activity, physical inactivity, nutrition and self-esteem. The influence of the primary care-giver on the children's physical activity and nutritional behaviors may lead to greater or lesser rates of obesity in childhood and eventually lead to adult obesity. Therefore, the intention of this intervention is to educate primary care-givers so as to effect change (in a positive way) in the children they care for. Assessment on steps taken, BMI, percent body fat, diet, self reported physical activity and diet will be used to evaluate the impact of the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Currently having a third grader attending public school

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2004-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | 3 years

SECONDARY OUTCOMES:
steps | 3 years
Percent body fat | 3 years
Basal metabolic rate | 3 years
Diet information (child and primary care-giver) | 3 years
Physical Activity and Inactivity information (child and primary care-giver) | 3 years
Self esteem measures | 3 years
Knowledge and attitudes | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mozhdeh B Bruss, PhD, Principal Investigator — Western Michigan University
Locations (1):
- Commonwealth of the Northern Mariana Islands Public School System, Saipan, Northern Mariana Islands